CLINICAL TRIAL: NCT04683068
Title: A Randomized Controlled Trial Comparing Self-referred Message to Family-referred Message Promoting Men's Adherence to Evidence-based Guidelines on BRCA1/2 Germline Genetic Testing: a Study Protocol
Brief Title: Promoting Men's Adherence to BRCA1/2 Germline Genetic Testing
Acronym: BRCA-MEN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: R1249/20-IEO1314
Record Dates: First submitted 2020-12-21; First posted 2020-12-24 (Actual); Last update posted 2022-05-13 (Actual); Status verified 2022-05

CONDITIONS: BRCA1 Mutation; BRCA2 Mutation; Psychosocial Factors

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- First-person gain-framed self-referred messages (Active Comparator): This group receives a message in which the main character is a man who speaks in first-person. The character is a man with a sister with a BRCA germline mutation. After this common introduction, the content of the messages becomes different.
  Group 1 receives a self-referred narrative message in which the protagonist explains that he has decided to have a genetic test to discover BRCA germline mutation. He then explains the reasons why this decision is important to himself (e.g., implementing preventive behaviors) and what are the possible benefits for the individual.
  Interventions: Behavioral: Message comparison
- First-person gain-framed family-referred messages (Experimental): This group receives a message in which the main character is a man who speaks in first-person. The character is a man with a sister with a BRCA germline mutation. After this common introduction, the content of the messages becomes different.
  Group 2 receives a family-referred narrative message in which the frame is similar to the previous message, but the character this time explains what are that the benefits for his family and why his decision to have a genetic test is important to them.
  Interventions: Behavioral: Message comparison

INTERVENTIONS:
Behavioral: Message comparison — Message comparison

SUMMARY:
BRCA1- and BRCA2-associated Hereditary Breast and Ovarian Cancer Syndrome (HBOC) increases the relative and absolute risk of developing breast and ovarian cancer and, to a lesser extent, prostate and pancreatic cancer. Men face BRCA-related cancer risks as women do, although with a different magnitude, and they may also transmit the mutations to their children. Notwithstanding, men have not received much attention since now. They are under-tested compared to women and the communication is not tailored on their needs. Research on the psychological determinants of men's informed decision-making is particularly lacking as well as experimental evidence on the efficacy of tailored messages on men's needs. Applying principles of the Health Action Process Approach (HAPA), the present protocol proposes a study with the aim to test psychological variables influencing men's decision-making. Moreover, the proposed research intends to test the efficacy of two messages through a randomized experimental study. A total of 264 participants will be involved, among the men's relatives of women with verified germline mutations. The study entails a pre- post- evaluation with randomization of the participants in two conditions corresponding to the two messages. The expected results provide answers related to the impact of action self-efficacy, outcome expectancy (personal or familiar), risk perception, health risk aversion, intolerance of uncertainty, perceived barriers, and coping self-efficacy on informed decision-making. Data gathered from this study may inform health care providers, policymakers, and public health managers about the communication strategy for men and about the psychological variables influencing decision-making.

DETAILED DESCRIPTION:
Background As for other pathogenic gene mutations [1,2], germline mutations in BRCA1- and BRCA2 genes (BReast CAncer 1 gene and BReast CAncer 2 gene) predispose carriers to an increased suscepti-bility in developing breast and ovarian cancer [3] but also prostate, pancreatic cancer and mela-noma [4]. BRCA1 and BRCA2 germline mutations are inherited in an autosomal dominant manner; this means that offspring of an individual with a BRCA1 or BRCA2 germline mutation have a 50% chance of inheriting the variant [5,6], and the same probability of passing it to the progeny. BRCA1/2 mutations have no gender distinction [7], both men and women can inherit the mutation, although it exposes them to different risks.

Men with BRCA1/2 mutations can incur a lifetime risk of up to 6.8 percent for breast cancer, and between 6 and 15 percent for prostate cancer [6,8]. These risks are particularly higher when BRCA2 gene is involved. However, men do not receive the same attention as women [9]. In particular, women can be tested to search BRCA1 or BRCA2 unknown germline mutations, especially when suffering from breast and/or ovarian cancer, or to search known BRCA1/2 germline mutations previously identified in the family (i.e., cascade screening). Instead, men are mainly involved in cascade screening and, rarely, they are tested for BRCA1/2 germline mutations [10]. Very recently, the guidelines of the National Comprehensive Cancer Network [11] have suggested to con-sider patients with pancreatic and prostatic cancers as eligible for genetic testing for BRCA germline mutations. However, such a recommendation is not yet routine for the test proposal.

Some socio-cultural aspects have been related to the men's attitude toward BRCA1/2 mutations and genetic testing. For example, Pritchard [12] suggested that BRCA 1/2 mutations are generally associated with female gender. He also pointed out that the name of the associated Hereditary Breast and Ovarian Cancer Syndrome (HBOC) creates a confusion since breast and ovarian cancers are considered a 'female matter' by layperson [18]. Similarly, others [13,14] have found that fear of stigmatization is one obstacle for the men's decision-making. To date, there are no studies, applying a strong theoretical rationale, that have systematically tested which are the psychological variables influencing men's informed decisions for genetic testing, when facing BRCA-related mutations. Moreover, to the best of our knowledge, there are no studies testing what is the better communication strategy to inform men's decision-making. Therefore, the present study aims to fill these gaps with an experimental study with a longitudinal component. First, applying principles of the Health Action Process Approach (HAPA), a motivational inclined theory that explains changes in behaviors, will be tested what psychological determinants influence the decision to undergo a genetic test for a germline BRCA mutations. The role of intolerance to the uncertainty and the health risk attitudes will be explored. The HAPA model has been chosen because it is an evolution of the first stadial models of health psychology [15] and it assumes that individuals pass through qualitatively different stages of psychological elaboration when they have to adopt new health behaviors. The other aim the proposed study is to test two different narrative messages in order to understand which is the most efficient in informing men's decision-making.

Principles of the Health Action Process Approach (HAPA) According to the Health Action Process Approach [16] there are several variables involved in the implementation of new health behaviors. Specifically, it is possible to identify risk perception, outcome expectancies and action self-efficacy as predisposing factors that have an impact on the informed decision; this is considered the motivation phase, in which subjects begin to form an intention. In this model, the intention to perform a specific health behavior is considered as a middle-level mediator between the variables considered in the motivation phase and those in the volition phase.

Furthermore, according to this model, volition factors involve planning that is further specified as coping and action planning, and coping self-efficacy. Volition factors are considered as be-ing influential in the subsequent phase and they are the most proximal predictors to actual behavior decisions. This second phase (i.e., the volition phase) should be subdivided in pre-action phase, in which the previous mentioned coping and action planning, and coping self-efficacy take place, and action phase, ending with a behavior.

This model was tested in several health contexts [17,18], in particular for smoking behavior [16,19,20], physical activity [21,22], dietary [23,24] and also in cancer-related screening behavior [25]. Those studies demonstrated the efficacy of the theory in explaining the initiation and maintenance of such health preventive behaviors. Together with the principles of the HAPA model, the present study aims to understand whether other psychological factors may explain men's decision making regarding genetic testing for BRCA1/2 germline mutations. For this reason, two attitudinal factors are examined: intolerance of uncertainty and health risk attitudes.

When people face with a potential threat for their health, one key element affecting their subsequent decisions and behaviors is how much they feel certain or uncertain regarding the threat. In our case, a man who is considering the possibility to undergo a genetic test for BRCA germline mutations is facing with two different types of uncertainty. The first one is the proximal uncertain-ty due to the result of the genetic test itself. The second one is the distal uncertainty depending on the risk to develop a cancer if a germline mutation would be found. The intention to undergo a genetic test for a germline mutation may be, therefore, determined by the way in which the individual manages the uncertainty due to the discovery of a possible negative result (i.e., the presence of a mutation) and to the future consequences of the germline mutation.

Intolerance of Uncertainty (IU) is a trait characteristic of individuals who are not able to tolerate the aversive reactions triggered by a perceived lack of sufficient information or by an is-sue that can have more than one solution [26]. Individuals with low tolerance for uncertainty tend to perceive the threat as a source of discomfort and to react negatively to it [27]. Some studies investigated the relationship between intolerance of uncertainty (IU) and the attitude to undergo health monitoring, in particular cancer-related screening [28,29]. In particular Tan and colleagues showed that intolerance of uncertainty may function as an important determinant of anxiety among men pursuing active surveillance for prostate cancer [28]. One qualitative study in lung cancer screening decision-making showed that some participants sought to decrease uncertainty through lung cancer screening and, if needed, with additional testing; others declined the screening in order to avoid the uncertainty associated with undefined results [30]. Indeed intolerance of uncertainty consists of two dimensions: the first one, the desire for predictability, is an active strategy to manage the uncertainty that is perceived as intolerable, and leads to search for as much information as possible about the threat to restore a balance. Rosen and colleagues [31] showed that high levels of IU were associated with an increase in health monitoring and screening; other studies suggested that searching for threat-related information may be driven by the desire to reduce uncertainty [32,33]. The second one, called uncertainty paralysis, is configured as an avoidance strategy and leads to inability to act because of the uncertainty [26].

Another construct related to the previous one, at least in the health framework, is the attitude toward health risk. In order to contrast the perception of significant uncertainty, people choose responses and act in a certain way, and this is defined as the personal attitude toward health risk. In fact, people differ in their attitude towards health risks, and this affects decision making regarding preventive behaviors (e.g., screening, physical activity), and risky behaviors (e.g., surgery) [34]. Taken together all this evidence suggest that IU and health risk attitudes may play a role when a man is facing with the decision to undergo a genetic test to detect BRCA germline mutation because there are similar mutations in the family. Since men with BRCA-related cancer risks deal with probabilistic and complex information [35,36], both of these attitudinal factors can have an effect on the implementation of health behaviors and therefore can influence the informed decision to undergo cascade screening for BRCA1/2 mutations.

How to inform men's decision making for BRCA1/2 germline mutations genetic testing The other aim is to investigate how to inform men's decision-making. Low levels of men's knowledge regarding BRCA1/2 germline mutations is found as one of the most important problems in this field [37]. Therefore, one main research achievement may be to find the right way to correctly inform them. The present study aims to test two different messages tailored to men's specific needs and to understand what is the best way to inform them. Although narrative approaches showed efficacy in promoting health behavioral intentions [38], and in increasing adherence to cancer screening [39] in particular, its utility for improving men's BRCA cascade screen-ing remains unexplored. The present research intends to explore whether narrative messages can be effective in informing men's decision-making.

In particular, two features are fundamental in narrative strategies context: the narrative perspective and the framing. The first one is a fundamental story feature and changes how information is delivered to the audience; researchers identified that first-person narrative messages are able to increase self-identity and to promote the assimilation of the theme better than third-person narratives [40]. Therefore, the present study chooses to create narrative messages with a first-person feature. Regarding the framing, messages can either emphasize negative consequences (losses) or positive outcomes (gains) of a given action. Prospect theory [41] posits that, in general, people are more likely to take risks when presented with a loss-framed message, and the contrary for a gain-framed message. But regarding disease prevention behaviors, like smoking cessation [61] and skin cancer prevention [42], researchers have suggested an advantage, albeit small, of a gain frame over a loss frame [43]. Therefore, the present study chooses to create narrative messages oriented to a gain frame.

Furthermore, applying the Uncertainty Management Theory [44], a social psychological approach to uncertainty, Rauscher et al. [13] investigated how men with increased BRCA-related cancer risk approach the individual and familial uncertainty related to that pathogenic variant. Those qualitative results showed that men's primary concern when managing BRCA-related cancer risks is the aversive consequences of the discovery of a germline mutation for their family [45]. Their focus on familial uncertainty management is maybe due to the difficulties encountered in the management of their own risk due to the lack of information and management options. In the end, the authors suggested that genetic counseling would benefit from a family focus. Also Hallowell and colleagues [46] highlighted the role of family member (mother, partner or children) in men's decision-making about BRCA testing. In particular, they showed how men's decision to have genetic testing was influenced by the obligations perceived from family members, primarily their children.

Based on these premises, this study proposes to test the effectiveness of two first-person gain-framed messages, one narrating a self-referred story and the other a family-referred story. The effectiveness will be measured in terms of one or both messages' ability to predict the intention to undergo genetic screening.

Objectives

We hypothesize the following relationships (figure 1 shows the tested model):

1. HP1: higher risk perception, positive outcome expectations, and action self-efficacy longitudinally predict the intention and the action to undergo a genetic test for BRCA germline mutations.
2. HP2: higher health risk attitude and low intolerance to uncertainty have a longitudinal influence on predicted higher intention, planning, and action initiation.
3. HP3: higher intention and coping self-efficacy longitudinally predict higher planning.
4. HP4: higher planning (i.e., action planning, coping planning) and coping self-efficacy longitudinally predict higher action initiation.
5. Based on results by Rauscher et al. [13] and Hallowell and colleagues [46], we formulated a research question: (RQ1) is there any difference between personal outcome expectations and family outcome expectations in their association with intention?
6. HP5: family-referred narrative gain-framed message (vs. self-referred narrative gain-framed message) will produce greater intention and action to undergo genetic testing for BRCA 1/2 germline mutations in at-risk men.

   Method Design The research will involve three phases, with results from each phase informing the next phase (see Figure 2). In the first phase, a literature review will be performed to identify other psychological variables influencing individuals' adherence to evidence based guidelines on BRCA1/2 germline genetic testing. Subsequently, a pilot survey will be created in order to test its feasibility and un-derstandability for participants.

   The third and final phase entails a RCT with participants receiving one of the two conditions (i.e., self-referred narrative framed message, family-referred narrative framed message) and it tests the main hypotheses and research question of the study. Participants will answer to several questions before and after the message exposure.

   Participants and study setting Participants are 264 males, relatives of women with BRCA1 and/or BRCA2 germline mutations who are patients of the Division of Cancer Prevention and Genetics at the European Institute of Oncology (IEO) in Milan. The IEO is a specialized Hospital and an internationally recognized Cancer Center located in Italy working on research, prevention, diagnosis, and treatment of cancer.

   Sample size and power calculation The sample size is determined through an a priori power analysis using GPower 4.0 [47]. Among the imputed parameters it was chosen to include partial η2 = .05, alpha lower than .05, power d (1-B) = .70. Considering that Luszczynska et al. [48] found a η2 = .01, η2 = .05 is a prudential choice. Two groups, corresponding to the two experimental conditions of the study, and 7 covariates were included. The final estimated number of participants is 264, 132 in each group. It should be noted that changing the number of covariates does not change the total number of participants.

   Recruitment According to the registry of the Division of Cancer Prevention and Genetics (IEO), all women with BRCA1 and/or BRCA2 germline mutations with at least a male relative will be reached by a phone call and/or an email. During the first contact, a member of the research team informs the female patients about the research purposes and the procedure. The researcher will then ask the women to share the information with their male relative(s) and to invite him (them) to participate in the research. All the information about the research, including an invitation letter, an information sheet, and the consent form, will be also sent by email to the women. If those relatives want to be contacted to participate in the study, a researcher calls them and shares with them the information sheet, the informed consent, and the link to the online survey. Participants will sign the informed consent before starting to fill the survey and data collection will be done through an online survey via the use of an identifier. In order to promote participant retention and complete follow-up, participants will be prompted to respond, calling them by phone or contacting them by email.

   Randomization Participants who meet the study inclusion criteria will be randomly assigned to receive one of the two conditions. Randomization will occur during T1, immediately after the data collection of psychological measures. The participants will not be informed of the condition to which they have been allocated until the message itself will be shown.

   Time 1 assessment All participants will complete the T1 assessment, via an online survey which will be available for a two-week period. The T1 measures will include demographic, health status, risk perception, health risk aversion, and intolerance of uncertainty. After this evaluation, participants will be ran-domized and exposed to one message. A manipulation check, the evaluation of the perceived qual-ity of the information presented on the messages, positive outcome expectations, action self-efficacy, benefit for genetic test will be then collected.

   Intervention Time 2 assessment Two weeks later, via an online survey, participants reply to questions on the intention to undergo germline genetic testing, coping self-efficacy, action planning, and coping planning.

   Time 3 assessment Starting from the end of T2 until 3 months later, data on action initiation will be collected (i.e., genet-ic test for BRCA1/2 gene germline mutations).

   Measures T1 measures Before the randomization, all participants answer several questions, as follows.

   Demographic. Self-reported age, education, occupation, degree of relationship with the woman with BRCA1/2 genes germline mutation, household composition.

   Health Status. Self-reported general health and existing diagnosis for the chronic disease will be investigated with a single item each [49]. Response options for general health conditions will be on a 5-point Likert scale. The response options for the item on the existing chronic disease will be binary coded (no - yes, specify).

   Risk perception. Relative risk perception regarding the possibility to develop breast, prostatic, and pancreatic cancer will be investigated with one item each [50,51]. Response options are on a 7-point Likert scale.

   Health Risk aversion. The six items of the Health Risk Attitude [52] will be administered to assess how a person would resolve risky health decisions. Response options are on a 7-point Likert scale.

   Intolerance of Uncertainty. The items of the Intolerance of Uncertainty Scale-12 [53] will be applied to measure two dimensions of the intolerance of ambiguity, which are the desire of predictability and uncertainty paralysis. Response options are on a 5-point Likert scale.

   T2 measures After the message exposure, participants reply to several questions, as follows.

   Manipulation check. Two items created ad hoc evaluate whether participants have read and understood the message content. Multiple-choice answers are used with one correct answer and two incorrect answers as distractors. Participants who fail to answer those questions will be excluded from the analyses.

   Perceived Quality of the Message. Three items evaluate whether the message is credible, convincing, and persuasive. Response options are on a 7-point Likert scale.

   Positive Outcome Expectation. Eight items will be created ad hoc for this research evaluating positive outcome expectations regarding the participant himself (4 items) and his family members (4 items). The response option will be on a 5-point Likert scale.

   Action Self-Efficacy. According to Schwarzer & Luszczynska's [16] indications, self-efficacy will be assessed through three items as the capability of keeping up with the behavior, by implementing coping strategies. Response option will be on a 5-point Likert scale.

   Benefit for Genetic Test. A 5-digit semantic differential will be applied to measure the perceived benefit for genetic tests. Examples of the proposed adjectives are important, relevant, useful, benefit.

   Intention to undergo genetic testing. Coping Self-efficacy. Three items created ad hoc for the present research evaluate whether the individual feels to be capable of tackling the possible obstacles and difficulties that could make it difficult to undergo genetic screening. Response options are on a 5-point Likert scale.

   Action planning. Three items developed ad hoc for the present research will ask if the participant has planned when, how, and where to undergo the genetic test for BRCA1/2 mutations. The response option will be on a 4-point Likert scale.

   Coping Planning. Four items developed ad hoc for the present research will ask how much the participant thinks to encounter in planning the action. The response option will be on a 5-point Likert scale.

   T3 measures Action. Information on the action initiation (i.e., a genetic test for BRCA1/2 germline mutations) will be collected when the participant takes the appointment for the genetic test and receives the test.

   References
   1. Corso G, Montagna G, Figueiredo J, Vecchia C La, Romario UF, Fernandes MS, et al. Heredi-tary gastric and breast cancer syndromes related to CDH1 germline mutation: A multidisciplinary clinical review. Cancers (Basel). MDPI AG; 2020. p. 1-25.
   2. Corso G, Bonanni B, Veronesi P, Galimberti V. Mutual exclusion of CDH1 and BRCA germline mutations in the pathway of hereditary breast cancer. Arch. Gynecol. Obstet. Springer Verlag; 2018. p. 1067-8.
   3. Corso G, Feroce I, Intra M, Toesca A, Magnoni F, Sargenti M, et al. BRCA1/2 germline mis-sense mutations: A systematic review. Eur. J. Cancer Prev. Lippincott Williams and Wilkins; 2018. p. 279-86.
   4. Nyberg T, Frost D, Barrowdale D, Evans DG, Bancroft E, Adlard J, et al. Prostate Cancer Risks for Male BRCA1 and BRCA2 Mutation Carriers: A Prospective Cohort Study. Eur Urol. Elsevier B.V.; 2020;77:24-35.
   5. Kuchenbaecker KB, Hopper JL, Barnes DR, Phillips KA, Mooij TM, Roos-Blom MJ, et al. Risks of breast, ovarian, and contralateral breast cancer for BRCA1 and BRCA2 mutation carriers. JAMA - J Am Med Assoc. American Medical Association; 2017;317:2402-16.
   6. Petrucelli N, Daly MB, Pal T. BRCA1- and BRCA2-Associated Hereditary Breast and Ovarian Cancer. GeneReviews®. University of Washington, Seattle; 1993.
   7. Silvestri V, Leslie G, Barnes DR, Agnarsson BA, Aittomäki K, Alducci E, et al. Characteriza-tion of the Cancer Spectrum in Men with Germline BRCA1 and BRCA2 Pathogenic Variants: Re-sults from the Consortium of Investigators of Modifiers of BRCA1/2 (CIMBA). JAMA Oncol. American Medical Association; 2020;6.
   8. Oh M, Alkhushaym N, Fallatah S, Althagafi A, Aljadeed R, Alsowaida Y, et al. The association of BRCA1 and BRCA2 mutations with prostate cancer risk, frequency, and mortality: A meta-analysis. Prostate. John Wiley and Sons Inc.; 2019;79:880-95.
   9. da Silva TL. Male breast cancer: Medical and psychological management in comparison to fe-male breast cancer. A review. Cancer Treat. Commun. Elsevier Ltd; 2016. p. 23-34.
   10. Marabelli M, Calvello M, Bonanni B. Test more men for BRCA genes. Nature. 2019;573:346.
   11. Daly MB, Pilarski R, Yurgelun MB, Berry MP, Buys SS, Dickson P, et al. Genetic/familial high-risk assessment: Breast, ovarian, and pancreatic, version 1.2020 featured updates to the NCCN guidelines. JNCCN J Natl Compr Cancer Netw. Harborside Press; 2020;18:380-91.
   12. Pritchard CC. New name for breast-cancer syndrome could help to save lives. Nature. Nature Research; 2019. p. 27-9.
   13. Rauscher EA, Dean M, Campbell-Salome G, Barbour JB. "How do we rally around the one who was positive?" Familial uncertainty management in the context of men managing BRCA-related cancer risks. Soc Sci Med. Elsevier Ltd; 2019;242:112592.
   14. Strømsvik N, Råheim M, Yen N, Gjengedal E. Men in the women's world of hereditary breast and ovarian cancer-a systematic review. Fam Cancer. Springer; 2009;8:221-9.
   15. Prochaska JO, Di Clemente CC. Transtheoretical therapy: Toward a more integrative model of change. Psychotherapy. American Psychological Association (APA); 1982;19:276-88.
   16. Schwarzer R, Luszczynska & A. The Health Action Process Approach. Eur Psychol. 2008;13:141-51.
   17. Zhang CQ, Zhang R, Schwarzer R, Hagger MS. A Meta-Analysis of the Health Action Process Approach. Heal Psychol. 2019;
   18. Mohammadi Zeidi I, morshedi H, shokohi abdolah. Application of the Health Action Process Approach (HAPA) Model to Determine Factors Affecting Physical Activity in Hypertensive Pa-tients. J Jiroft Univ Med Sci. Journal of Jiroft University of Medical Sciences; 2020;7:349-60.
   19. Radtke T, Scholz U, Keller R, Hornung R. Smoking is ok as long as I eat healthily: Compensa-tory Health Beliefs and their role for intentions and smoking within the Health Action Process Ap-proach. Psychol Heal. 2012;27:91-107.
   20. Scholz U, Nagy G, Göhner W, Luszczynska A, Kliegel M. Changes in self-regulatory cogni-tions as predictors of changes in smoking and nutrition behaviour. Psychol Heal. 2009;24:545-61.
   21. Barg CJ, Latimer AE, Pomery EA, Rivers SE, Rench TA, Prapavessis H, et al. Examining pre-dictors of physical activity among inactive middle-aged women: An application of the health ac-tion process approach. Psychol Heal. Routledge ; 2012;27:829-45.
   22. Parschau L, Barz M, Richert J, Knoll N, Lippke S, Schwarzer R. Physical activity among adults with obesity: Testing the health action process approach. Rehabil Psychol. American Psychologi-cal Association Inc.; 2014;59:42-9.
   23. Steca P, Pancani L, Greco A, D'Addario M, Magrin ME, Miglioretti M, et al. Changes in Die-tary Behavior among Coronary and Hypertensive Patients: A Longitudinal Investigation Using the Health Action Process Approach. Appl Psychol Heal Well-Being. Wiley-Blackwell; 2015;7:316-39.
   24. Chiu C-Y, Lynch RT, Chan F, Rose L. The Health Action Process Approach as a Motivational Model of Dietary Self-Management for People With Multiple Sclerosis. Rehabil Couns Bull. SAGE PublicationsSage CA: Los Angeles, CA; 2012;56:48-61.
   25. Daniel AO, Omorogieva Enoma I, Omobude-Idiado SN. Application of Protection Motivation Theory (PMT) and Health Action Process Approach (HAPA) in promoting women's adaptive en-gagement towards breast self examination. Acad Res Int. 2014;5:291.
   26. Carleton RN. Fear of the unknown: One fear to rule them all? J. Anxiety Disord. Elsevier Ltd; 2016. p. 5-21.
   27. Buhr K, Dugas MJ. Investigating the construct validity of intolerance of uncertainty and its unique relationship with worry. J Anxiety Disord. J Anxiety Disord; 2006;20:222-36.
   28. Tan H-J, Marks LS, Hoyt MA, Kwan L, Filson CP, Macairan M, et al. The Relationship be-tween Intolerance of Uncertainty and Anxiety in Men on Active Surveillance for Prostate Cancer. J Urol. Elsevier Inc.; 2016;195:1724-30.
   29. Taber JM, Klein WMP, Ferrer RA, Han PKJ, Lewis KL, Biesecker LG, et al. Perceived ambi-guity as a barrier to intentions to learn genome sequencing results. J Behav Med. Springer New York LLC; 2015;38:715-26.
   30. Schapira MM, Aggarwal C, Akers S, Aysola J, Imbert D, Langer C, et al. How patients view lung cancer screening: The role of uncertainty in medical decision making. Ann Am Thorac Soc. American Thoracic Society; 2016;13:1969-76.
   31. Rosen NO, Knäuper B, Sammut J. Do individual differences in intolerance of uncertainty af-fect health monitoring? Psychol Heal. Routledge ; 2007;22:413-30.
   32. Hock M, Krohne HW, Kaiser J. Coping Dispositions and the Processing of Ambiguous Stimuli. J Pers Soc Psychol. American Psychological Association Inc.; 1996;70:1052-66.
   33. Krohne HW. Vigilance and cognitive avoidance as concepts in coping research. Atten Avoid Strateg coping with aversiveness. 1993.
   34. Van Osch SMC, Stiggelbout AM. The development of the Health-Risk Attitude Scale. 2007.
   35. Oliveri S, Pravettoni G. Capturing how individuals perceive genetic risk information: a phe-nomenological perspective. J Risk Res. Routledge; 2018;21:259-67.
   36. Oliveri S, Scotto L, Ongaro G, Triberti S, Guiddi P, Pravettoni G. "You do not get cancer by chance": Communicating the role of environmental causes in cancer diseases and the risk of a "guilt rhetoric." Psychooncology. John Wiley and Sons Ltd; 2019;28:2422-4.
   37. Skop M, Lorentz J, Jassi M, Vesprini D, Einstein G. "Guys Don't Have Breasts": The Lived Experience of Men Who Have BRCA Gene Mutations and Are at Risk for Male Breast Cancer. Am J Mens Health. SAGE Publications Inc.; 2018;12:961-72.
   38. Braddock K, Dillard JP. Meta-analytic evidence for the persuasive effect of narratives on be-liefs, attitudes, intentions, and behaviors. Commun Monogr. Routledge; 2016;83:446-67.
   39. Jensen JD, King AJ, Carcioppolo N, Krakow M, Samadder NJ, Morgan S. Comparing tailored and narrative worksite interventions at increasing colonoscopy adherence in adults 50-75: A ran-domized controlled trial. Soc Sci Med. 2014;104:31-40.
   40. van Peer W, Maat HP. Narrative perspective and the interpretation of characters' motives. Lang Lit Int J Stylist. SAGE Publications Ltd; 2001;10:229-41.
   41. Kahneman D, Tversky A. Prospect Theory: An Analysis of Decision Under Risk. 2013. p. 99-127.
   42. O'Keefe DJ, Jensen JD. The relative persuasiveness of gain-framed and loss-framed messages for encouraging disease prevention behaviors: A meta-analytic review. J. Health Commun. Taylor & Francis Group ; 2007. p. 623-44.
   43. Kim HK, Lee TK. Conditional Effects of Gain-Loss-Framed Narratives among Current Smok-ers at Different Stages of Change. J Health Commun. Taylor and Francis Inc.; 2017;22:990-8.
   44. Brashers DE. Communication and Uncertainty Management. J Commun. Oxford University Press (OUP); 2001;51:477-97.
   45. Hesse-Biber S, An C. Within-Gender Differences in Medical Decision Making Among Male Carriers of the BRCA Genetic Mutation for Hereditary Breast Cancer. Am J Mens Health. SAGE Publications Inc.; 2017;11:1444-59.
   46. Hallowell N, Ardern-Jones A, Eeles R, Foster C, Lucassen A, Moynihan C, et al. Men's Deci-sion-Making About Predictive BRCA1/2 Testing: The Role of Family. J Genet Couns. John Wiley & Sons, Ltd; 2005;14:207-17.
   47. Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: A flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. Psychonomic Society Inc.; 2007. p. 175-91.
   48. Luszczynska A, Schwarzer R, Lippke S, Mazurkiewicz M. Self-efficacy as a moderator of the planning-behaviour relationship in interventions designed to promote physical activity. Psychol Heal. Psychol Health; 2011;26:151-66.
   49. Shim M, Kelly B, Hornik R. Cancer information scanning and seeking behavior is associated with knowledge, lifestyle choices, and screening. J Health Commun. J Health Commun; 2006;11:157-72.
   50. Renner B. Hindsight bias after receiving self-relevant health risk information: A motivational perspective. Memory. Taylor & Francis Group ; 2003;11:455-72.
   51. Renner B. Biased Reasoning: Adaptive Responses to Health Risk Feedback. Personal Soc Psy-chol Bull. Pers Soc Psychol Bull; 2004;30:384-96.
   52. Dieteren CM, Brouwer WBF, Van Exel J. How do combinations of unhealthy behaviors relate to attitudinal factors and subjective health among the adult population in the Netherlands? BMC Public Health. BioMed Central Ltd.; 2020;20:441.
   53. Bottesi G, Ghisi M, Novara C, Bertocchi J, e Ilaria MB, Dominicis D, et al. Intolerance of un-certainty scale (IUS-27 e IUS-12): Due studi preliminari. Psicoter Cogn e Comport. 2015;21:345-65.

ELIGIBILITY:
Inclusion Criteria:

* Male relatives of patients with an established germline genetic mutation (pathogenic or likely pathogenic variants) of the BRCA1 and / or BRCA2 genes
* Aged ≥ 18
* Able to give informed consent
* Able to read, speak, and understand Italian

Exclusion Criteria:

* BRCA1 and / or BRCA2 germline genetic screening load detected
* Diagnosis of breast, pancreatic, or prostate cancer

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 264 (Actual)
Dates: Start 2021-01-10 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Intention to undergo genetic testing | 2-3 weeks after the intervention exposure
  The intention of undergoing genetic testing is measured through three items evaluating the urge to engage the behavior. Example of item is: "In the next few months, do you have the intention of planning a genetic screening?". Response options are on a 5-point Likert scale.

SECONDARY OUTCOMES:
Action | Until 3 months after the intervention exposure
  Information on the action initiation (i.e., genetic test for BRCA1/2 germline mutations) will be col-lected when the participant takes the appointment for the genetic test and receives the test.

CONTACTS AND LOCATIONS:
Overall Officials: Serena Petrocchi, Principal Investigator — European Institute of Oncology
Locations (1):
- European Institute of Onocolgy, Milan, MI, Italy

REFERENCES:
- [Derived] Petrocchi S, Ongaro G, Calvello M, Feroce I, Bonanni B, Pravettoni G. A randomized controlled trial comparing self-referred message to family-referred message promoting men's adherence to evidence-based guidelines on BRCA1/2 germline genetic testing: A registered study protocol. PLoS One. 2022 Apr 8;17(4):e0266327. doi: 10.1371/journal.pone.0266327. eCollection 2022. PMID 35395021